CLINICAL TRIAL: NCT03864380
Title: Analysis of the Variation of the Retinal Vascularization After a Prolonged Effort
Acronym: MARETINE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2018_10
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Retinal Vascular Disorder; Sport Injury
Keywords: Retinal Vascularization; Intense effort; OCT-A
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Person running a marathon: Exams performed before (1 month maximum) and after the marathon (1 hour maximum) :
  Color retinography Optical Coherence Tomography - Angiography (OCT-A) Blood pressure measurement
  Interventions: Diagnostic Test: Color retinography; Diagnostic Test: OCT-A; Diagnostic Test: Blood pressure measurement

INTERVENTIONS:
Diagnostic Test: Color retinography — Non mydriatic color retinography within 1 month before and within 1 hour after the marathon
Diagnostic Test: OCT-A — Optical Coherence Tomography - Angiography within 1 month before and within 1 hour after the marathon
Diagnostic Test: Blood pressure measurement — Blood pressure measurement within 1 month before and within 1 hour after the marathon

SUMMARY:
The cardiovascular parameters of prolonged physical exercice have been studied, but very little data is available about the retinal vascularization.

The eye allows in vivo visualization of micro-vascularisation and is considered as an excellent marker of general vascular condition.

The marathon is an intense and prolonged exercise (running 42.195 km) in aerobic environment. Thus the investigators propose to study the vascular parameters of the retina, before and after this physical exercise.

This will allow : 1) to collect information on the physiology of the retinal vascularization to prolonged effort, 2) to detect any retinal damage (haemorrhages, edema, occlusion ...), not known to date.

The results may highlight vascular effects related to retinal hypoxia (venous tortuosity, haemorrhage, venous occlusion, hypoxic edema). Furthermore the results may urge prevention in this sport more and more democratized.

the investigators hypothesized that prolonged physical exercice causes a change in retinal vascularization.

ELIGIBILITY:
Inclusion Criteria:

* Person registered at the 2019 Paris Marathon

Exclusion Criteria:

* Ophthalmological disorders making access to the fundus impossible for both eyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Person running a marathon
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Density of retinal vascular plexuses | up to 1 hour
  Percentage, Measurement with OCT-A

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mauget-Faysse M, Arej N, Paternoster M, Zuber K, Derrien S, Thevenin S, Alonso AS, Salviat F, Lafolie J, Vasseur V. Retinal and choroidal blood flow variations after an endurance exercise: A real-life pilot study at the Paris Marathon. J Sci Med Sport. 2021 Nov;24(11):1100-1104. doi: 10.1016/j.jsams.2021.03.013. Epub 2021 Mar 30. PMID 33824079